CLINICAL TRIAL: NCT05560776
Title: OPTimizing Endobronchial Ultrasound Sampling In Suspected Non Small Cell Lung Cancer for Molecular Markers : A Pragmatic Randomized Controlled TriaL
Brief Title: Optimizing Endobronchial Ultrasound Sampling for Molecular Markers for NSCLC
Acronym: OPTIMAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Principal Investigator, Marc Fortin, Primary investigator, Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-3850
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer; Circulating Tumor Cell
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Pathologist will be blinded to study arm when analyzing samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 passes per target on EBUS (Experimental)
  Interventions: Procedure: Endobronchial ultrasound
- 3 passes per target on EBUS (Experimental)
  Interventions: Procedure: Endobronchial ultrasound

INTERVENTIONS:
Procedure: Endobronchial ultrasound — Two or three passes per lymph node

SUMMARY:
In this monocentric randomized controlled trial, 120 potential non small cell lung cancer (NSCLC) patients for which tissue diagnosis and material for next generation sequencing (NGS) is required for clinical management will be approached the day of their endobronchial ultrasound to participate in the study. They will be randomized to 2 vs 3 passes/lymph node and will all undergo liquid biopsy. The co-primary outcomes are 1)the rate of obtention of adequate material for NGS testing with 2 vs 3 passes/lymph node and 2)the percentage of patients for which liquid biopsy allows to identify clinically pertinent findings not available from tissue biopsy

ELIGIBILITY:
Inclusion Criteria:

* Suspected or confirmed NSCLC requiring tissue sample for NGS testing to guide clinical management
* Presence of at least 2 targets accessible by EBUS or EUS suspicious of malignancy (primary tumor, lymph node > 10mm or with Standardized Uptake Value (SUV) > 2.5)

Exclusion Criteria:

* Other modality then EBUS judged preferable by treating physician to obtain tumoral tissue for NGS testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of obtention of adequate material for NGS testing with 2 vs 3 passes/lymph node | At recruitment completion (expected time 2 years), all cell blocks will be reviewed by the blinded pathologist to assess adequacy rate for NGS testing
  Cell block will be reviewed by a blinded pathologist to determine the percentage of tumor cells within the sample by increment of 5%. More than 10% of tumor cell will be considered adequate.
Percentage of patients for which liquid biopsy allowed to identify genetic alterations not identified from tissue biopsy | At 1 month
  A case for which liquid biopsy NGS testing allows to identify a genetic alteration not identified by matched tissue biopsy (tissue inadequate, insufficient for molecular testing or adequate but genetic alteration not found) will be considered a case for which liquid biopsy provided additional clinical findings

SECONDARY OUTCOMES:
Rate of obtention of adequate material for NGS testing with 2 vs 3 passes/patient | At recruitment completion (expected time 2 years), all cell blocks will be reviewed by the blinded pathologist to assess adequacy rate for NGS testing
  Cell block will be reviewed by a blinded pathologist to determine the percentage of tumor cells within the sample by increment of 5%. More than 10% of tumor cell will be considered adequate.
Rate of obtention of adequate material for NGS testing with 2 vs 3 passes/sampling scheme | At recruitment completion (expected time 2 years), all cell blocks will be reviewed by the blinded pathologist to assess adequacy rate for NGS testing
  Cell block will be reviewed by a blinded pathologist to determine the percentage of tumor cells within the sample by increment of 5%. More than 10% of tumor cell will be considered adequate.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fortin, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut Universitaire de Cardiologie et Pneumologie de Quebec, Québec, Quebec, Canada